CLINICAL TRIAL: NCT05547425
Title: WildCam: A Privacy Conscious Wearable Eating Detection Camera People Will Actually Wear in the Wild
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Nabil Alshurafa, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STU00213549; 1R03DK127128-01 (NIH)
Record Dates: First submitted 2022-05-24; First posted 2022-09-21 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Wearable Electronic Devices

STUDY DESIGN:
Intervention Model Description: Of the 3 obfuscation settings (blur, mask, cartoon), participants are randomly assigned to 1, which they test for the first or second 7-day test period. During the remaining test period, participants use WildCam with the raw images setting. There is a washout period between each test period. The order of the test sequence is counterbalanced across participants to reduce carryover effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Blur obfuscation (Experimental): Blurring is applied to objects and people in the background of images.
  Interventions: Device: Blur Obfuscation
- Edge obfuscation (Experimental): Objects and people in the background of images are replaced with an outline of the object.
  Interventions: Device: Edge Obfuscation
- Cartoon obfuscation (Experimental): Blurring is applied to objects and people in the background of images and the wearer's face is concealed with cartoon faces.
  Interventions: Device: Cartoon Obfuscation
- Raw images (Experimental): No editing is performed on images.
  Interventions: Device: Raw images

INTERVENTIONS:
Device: Blur Obfuscation — Blurring is applied to objects and people in the background of images.
  Arms: Blur obfuscation
Device: Edge Obfuscation — Objects and people in the background of images are replaced with an outline of the object.
  Arms: Edge obfuscation
Device: Cartoon Obfuscation — Blurring is applied to objects and people in the background of images and the wearer's face is concealed with cartoon faces.
  Arms: Cartoon obfuscation
Device: Raw images — No editing is performed on images.
  Arms: Raw images

SUMMARY:
WildCam is a wearable device that collects video data of the user's face and upper torso to capture eating behaviors. WildCam and its accompanying software is privacy conscious, meaning it utilizes a computer vision algorithm that extracts proximal features (the user's body and objects-in-hand) from the video and digitally obfuscates the distal features (background environment and entities therein) to preserve the privacy of the wearer, as well as any bystanders who may be in the device's visual field. The present study tests the impact of 3 different obfuscation techniques on acceptability, including the willingness of users to wear the device. Participants are randomly assigned to 1 of the 3 obfuscation techniques (blurring, masking, or cartooning). Participants wear the WildCam during waking hours during a 7-day period with the randomly selected obfuscation setting enabled and a 7-day period with the raw images (no obfuscation) setting. The order of these periods is counterbalanced, and the two periods are separated by a 7-day washout period during which WildCam is not worn. Structured feedback, including user burden and acceptability surveys, is collected to determine the efficacy of each obfuscation technique on increasing user acceptability, including willingness to use the WildCam device, as opposed to a video-collecting device without obfuscation.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30 or greater
* Chicago Metro Area resident
* Able to speak, read, and write in English
* Valid phone number
* Smartphone ownership
* Have Wi-Fi at home

Exclusion Criteria:

* 15% or greater weight change in last 3 months
* Medication related weight gain
* Genetic obesity syndrome (e.g., Prader-Willi, Bardet-Biedl, Cohen Syndrome)
* Member of household enrolled in study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Mean Wear Time | 7 days
  Average duration in minutes of data collected per day, calculated from video time stamps

SECONDARY OUTCOMES:
Acceptability | 7 days
  Score (0-80) obtained from User Burden Scale (Suh. et al 2016), collected post-study

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Department of Preventive Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No